CLINICAL TRIAL: NCT03931031
Title: Pre-surgical Evaluation for the Quantra System in Adult Patients Undergoing Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: HemoSonics LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: HEMCS-017
Record Dates: First submitted 2019-04-20; First posted 2019-04-29 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Blood Loss, Surgical
Keywords: Viscoelastic testing; Coagulation; Quantra; Hemostasis
MeSH Terms: conditions — Blood Loss, Surgical; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Cardiac Surgery Patients: Patients taking antiplatelet medication who are scheduled for elective cardiac surgery.
  Interventions: Diagnostic Test: Quantra System

INTERVENTIONS:
Diagnostic Test: Quantra System — Diagnostic device to monitor coagulation properties of a whole blood sample at the point-of-care
  Other Names: Quantra QPlus Cartridge

SUMMARY:
This study will evaluate the performance of the Quantra System comprised of the Quantra Hemostasis Analyzer with the QPlus Cartridge in patients taking anitplatelet medication that are scheduled to undergo cardiac surgery.

DETAILED DESCRIPTION:
The Quantra System is a fully integrated and automated in vitro diagnostic device which uses SEER Sonorheometry, an ultrasound-based technology, to characterize the viscoelastic properties of a whole blood sample during coagulation. The Quantra QPlus Cartridge was developed to monitor hemostasis during major surgical procedures in adult patients. The cartridge consists of four independent channels each containing different sets of reagents, which provide four measurements performed in parallel yielding six parameters that depict the functional status of a patient's coagulation system.

This single-site, prospective, observational study will evaluate the performance of the Quantra System as compared to standard coagulation tests and comparable measures determined using TEG in patients taking antiplatelet medication that are scheduled to undergo cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subject is scheduled for elective cardiac surgery utilizing cardiopulmonary bypass, including the placement of a ventricular assist device
* Subject was identified as taking antiplatelet medication, specifically a P2Y12 inhibitor such that a TEG Platelet Mapping test is prescribed prior to surgery to assess possible platelet inhibition
* Subject is ≥ 18 years
* Subject is willing to participate and he/she has signed a consent form

Exclusion Criteria:

* Subject is younger that 18 years
* Subject is unable to provide written informed consent
* Subject is incarcerated at the time of the study
* Subject is pregnant
* Subject is currently enrolled in a distinct study that might confound the results of the proposed study
* Subject is affected by a condition that, in the opinion of the clinical team, may pose additional risks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential study participants will be adult (≥ 18 years) subjects who are taking antiplatelet medication and who are scheduled for elective cardiac surgery utilizing cardiopulmonary bypass, including the placement of a ventricular assist device.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2020-04-07 (Actual); Study Completion 2020-06-27 (Actual)

PRIMARY OUTCOMES:
Comparison of Quantra Clot Time test results to TEG test results. | Prior to surgery (Baseline)
  Coagulation function assessed by Quantra and TEG.
Comparison of Quantra Clot Stiffness test results to TEG test results. | Prior to surgery (Baseline)
  Coagulation function assessed by Quantra and TEG.
Comparison of Quantra Clot Time and Clot Stiffness test results to TEG test results. | Post-bypass (10 to 20 minutes after protamine administration).
  Coagulation function assessed by Quantra and TEG.
Comparison of Quantra Clot Time test results to TEG test results. | Post-bypass (10 to 20 minutes after protamine administration).
  Coagulation function assessed by Quantra and TEG.
Comparison of Quantra Fibrinogen Contribution to Clot Stiffness test results to laboratory fibrinogen | Prior to surgery (Baseline)
  Coagulation function assessed by Quantra and laboratory fibrinogen testing
Comparison of Quantra Fibrinogen Contribution to Clot Stiffness test results to laboratory fibrinogen | Post-bypass (10 to 20 minutes after protamine administration).
  Coagulation function assessed by Quantra and laboratory fibrinogen testing
Comparison of Quantra Platelet Contribution to Clot Stiffness test results to laboratory platelet count | Post-bypass (10 to 20 minutes after protamine administration).
  Coagulation function assessed by Quantra and laboratory fibrinogen testing
Comparison of Quantra Platelet Contribution to Clot Stiffness test results to laboratory platelet count | Prior to surgery (Baseline)
  Coagulation function assessed by Quantra and platelet count

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsville Hospital, Huntsville, Alabama, United States

IPD SHARING:
Plan to Share IPD: No